CLINICAL TRIAL: NCT00001764
Title: Mycophenolate Mofetil in the Treatment of Wegener's Granulomatosis and Related Vasculitides
Brief Title: Mycophenolate Mofetil to Treat Wegener's Granulomatosis and Related Vascular Inflammatory Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980092; 98-I-0092
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-06

CONDITIONS: Vasculitis; Wegener's Granulomatosis
Keywords: Alternative agent; Purine Antimetabolite; Immunosuppressive; Previous relapse; Drug Intolerance; Wegener's Granulomatosis
MeSH Terms: conditions — Vasculitis; Granulomatosis with Polyangiitis | interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: Mycophenolate Mofetil

SUMMARY:
This study will examine the safety and effectiveness of the drug mycophenolate mofetil (MPM) in treating Wegener's granulomatosis and related inflammatory vessel diseases. Blood vessel inflammation in these patients may involve different parts of the body, including the brain, nerves, eyes, sinuses, lungs, kidneys, intestinal tract, skin, joints, heart, and other sites. The more severe the involvement, the more likely the disease will be life-threatening. Standard treatment consists of combination drug therapy with prednisone and a cytotoxic agent-usually cyclophosphamide or methotrexate. However, some patients in whom this treatment is initially successful have a disease relapse; other patients cannot take the medications because of other health problems or because of severe side effects of the drugs.

MPM is approved by the Food and Drug Administration to prevent kidney transplant rejection. It is chemically similar to another cytotoxic drug called azathioprine, which has been beneficial in maintaining remission in patients with Wegener's granulomatosis who have been treated successfully with cyclophosphamide. Because MPM is more effective than azathioprine in preventing organ rejection, it may also prove beneficial as a second-line treatment for Wegener's granulomatosis.

Patients with Wegener's granulomatosis or related inflammatory vessel diseases who have had a relapse following treatment with cyclophosphamide and methotrexate or who cannot take one or both of these drugs may be eligible for this study. Only patients who have been treated at NIH in the methotrexate protocol or the cyclophosphamide switching to methotrexate protocol, or who have received the exact same treatment from their own physician may participate.

Participants will have a complete medical evaluation including laboratory studies. Consultations, X-rays and biopsies of affected organs may also be done if indicated for diagnosis or treatment. Patients with active disease will be given MPM and prednisone, both in tablet form. Patients with inactive disease will receive only prednisone if they are already taking it. In both cases, the prednisone will be reduced gradually and discontinued if the disease improves significantly. MPM therapy will continue for at least 2 years. If after 2 years the disease remains in remission, the MPM dose will be gradually reduced and then stopped. If active disease recurs while on MPM therapy, the treatment plan will likely be changed. The new regimen will be determined by the severity of disease, other medical conditions, and history of side effects to previous medications.

Patients will be followed at the NIH clinic every month for the first 3 months on MPM and then every 3 months for another 18 months. Those whose disease has remained in remission and have stopped all medications will then be followed every 6 months for 4 visits. The follow-up visits will include a physical examination, blood draws, and, if needed, X-rays. Visits may be scheduled more frequently if medically indicated.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of mycophenolate mofetil in the treatment of Wegener's granulomatosis and related vasculitides in patients who have contraindications to methotrexate or cyclophosphamide or have experienced disease relapse while on these agents. Mycophenolate mofetil is a novel immunosuppressive agent which has been approved by the FDA for renal transplantation. It is chemically similar to and has a potentially greater efficacy in preventing acute transplant rejection than azathioprine, a drug which has been previously used as an alternative treatment for vasculitis. In this study, patients who have had disease relapse or contraindications to methotrexate will initially receive cyclophosphamide and glucocorticoids and then switch from cyclophosphamide to mycophenolate mofetil upon disease remission. If at the end of two years of mycophenolate mofetil therapy there is continued evidence of disease remission, the drug will be tapered and discontinued. Patients with contraindications to both cyclophosphamide and methotrexate will be treated initially with prednisone and mycophenolate mofetil with mycophenolate mofetil being continued for two full years after disease remission and then tapered and discontinued. For patients who develop intolerance to methotrexate or cyclophosphamide while their disease is in remission, mycophenolate mofetil will be started and continued for two years after which time it will be tapered and discontinued. Patients will be prospectively monitored for evidence of disease activity and drug toxicity. Specific parameters that will be obtained include the time to disease remission, the rate and time of disease relapse, and the incidence of drug related adverse effects.

ELIGIBILITY:
INCLUSION CRITERIA:

Documentation of Wegener's Granulomatosis (WG) based on clinical characteristics and histopathological evidence of vasculitis.

Patient with a positive C- or P-ANCA and glomerulonephritis as evidenced by the presence of red blood cell casts and proteinuria or renal biopsy showing necrotizing glomerulonephritis in the absence of positive immunofluorescence for immunoglobulin and complement will also be eligible.

Patients must be of the ages of 18-80 years.

Patients on the CYC to MTX protocol (#95-I-0091) who experience a relapse of disease while on MTX maintenance therapy. Relapse is defined by a Vasculitis Disease Activity Index of greater than or equal to 3. Patients from outside the NIH will also be eligible if they have been treated with a CYC to MTX regimen identical to that used in #95-I-0091 and experience a relapse of disease while on MTX maintenance therapy. If treatment for this relapse has already been commenced at the outside institution with daily CYC and glucocorticoid, patients will still be eligible if there is a history of a Vasculitis Disease Activity Index greater than or equal to 3 at the time of CYC and glucocorticoid initiation. Patients who experience a relapse of disease after MTX has been stopped or while tapering the MTX dose (following 2 years of maintenance therapy) will not be eligible.

Patients with active disease who have a contraindication to MTX therapy will be eligible. Evidence of active disease as defined by a Vasculitis Disease Activity Index of greater than or equal to 3.

Patients with inactive disease who have a contraindication to CYC and. Evidence of active disease as defined by a Vasculitis Disease Activity Index of greater than or equal to 3.

Patients with inactive disease on MTX while on the CYC to MTX protocol (95-I-0091) or the MTX protocol (90-I-0086) who develop an contraindication necessitating discontinuation of MTX. Patients from outside the NIH will also be eligible if they similarly develop a contraindication to MTX while on treatment.

Patients with inactive disease on the CYC protocol (#76-I-0041 or 76-I-0042) who develop a contraindication necessitating CYC discontinuation and also have a contraindication to receiving MTX. Patients from outside the NIH will also be eligible if they similarly develop a contraindication to CYC while on treatment and cannot receive MTX.

Patients with inactive disease who are receiving treatment with CYC and prednisone in a manner similar to #76-I-0042 will be eligible if they have a contraindication to receiving MTX and have been in remission for less 3 months.

EXCLUSION CRITERIA:

Evidence of active infection which, in the judgment of the investigator, is of greater danger to the patient than the underlying vasculitis. In those instances in which infection cannot be ruled out by gram stain and culture of secretions or collections of fluid in involved organs, it may be necessary to obtain a biopsy of the affected tissue for microbiological and histopathological studies.

Patients who are pregnant or who are nursing infants will not be eligible. Fertile women must have a negative pregnancy test within one week prior to study entry and must be using an effective means of birth control.

Patients with active disease who are eligible for the CYC to MTX protocol (#95-I-0091) or the MTX protocol (#90-I-0086).

Active peptic ulcer disease.

Serological evidence of infection with human immunodeficiency virus. A serological determination will be performed within two weeks of beginning study participation.

Inability to comply with study guidelines.

Creatinine clearance less than 25ml/min.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1998-04; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Simmons WD, Rayhill SC, Sollinger HW. Preliminary risk-benefit assessment of mycophenolate mofetil in transplant rejection. Drug Saf. 1997 Aug;17(2):75-92. doi: 10.2165/00002018-199717020-00001. PMID 9285199
- [Background] Fulton B, Markham A. Mycophenolate mofetil. A review of its pharmacodynamic and pharmacokinetic properties and clinical efficacy in renal transplantation. Drugs. 1996 Feb;51(2):278-98. doi: 10.2165/00003495-199651020-00007. PMID 8808168
- [Background] Goldblum R. Therapy of rheumatoid arthritis with mycophenolate mofetil. Clin Exp Rheumatol. 1993 Mar-Apr;11 Suppl 8:S117-9. PMID 8324935